CLINICAL TRIAL: NCT07196852
Title: Effects of N-acetylcysteine on Biological Responses to High-intensity Interval Training in Adults With Overweight/Obesity
Brief Title: Redox Status and Exercise Training-induced Adaptations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Dimitrios Draganidis, Assistant Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTH-2568_2.4.2025
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Overweight (BMI > 25); Obesity
Keywords: overweight; obesity; N-acetylcysteine; high-intensity interval training
MeSH Terms: conditions — Overweight; Obesity | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with repeated measures
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Experimental): Oral N-acetylcysteine supplementation for 12 weeks (2 x 600 mg capsules/day)
  Interventions: Dietary Supplement: N Acetyl L Cysteine
- Placebo (Placebo Comparator): Oral placebo supplementation for 12 weeks (2 placebo capsules/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: N Acetyl L Cysteine — Participants will participate in 3 multicomponent high-intensity interval training (m-HIIT) sessions per week over a 12-week period while receiving daily 1200 mg N-acetylcysteine (2 pills x 600 mg/day ).
  Arms: N-acetylcysteine
Dietary Supplement: Placebo — Participants will participate in 3 multicomponent high-intensity interval training (m-HIIT) sessions per week over a 12-week period while receiving daily 2 placebo pills/day.
  Arms: Placebo

SUMMARY:
Excess fat accumulation is a key feature of overweight and obesity that is mainly driven by nutrient overload and insufficient physical activity. White adipose tissue displays lipid overload and hypertrophy accompanied by macrophages infiltration, hypoxia, inflammation and excess production of reactive oxygen species (ROS). An inflammatory response and ROS production are also evident in other metabolism regulating tissues and organs such as skeletal muscle, liver, pancreas and hypothalamus, contributing to a chronic inflammatory state, redox status disturbances and metabolic complications. There is overwhelming evidence showing that adults with overweight/obesity exhibit lower glutathione (GSH) levels in blood erythrocytes, skeletal muscle cells and subcutaneous and visceral adipose tissue cells. GSH, a tripeptide consisting of the amino acids glutamate, cysteine and glycine, is the most abundant thiol-containing antioxidant in the human body and has been, recently, characterized as a novel therapeutic target for the treatment of numerous chronic diseases, due to its potent intracellular redox buffering capacity. Interestingly, lower GSH levels have been associated with diet-induced weight loss resistance, while enhancement of GSH levels through N-acetylcysteine (NAC) supplementation reduces markers of oxidative stress, inflammation, insulin resistance, hypertension, endothelia dysfunction and improves vitamin D metabolism. NAC is a thiol donor that elicits antioxidant effects by (i) directly scavenging ROS and (ii) providing reduced cysteine through deacetylation, which supports the biosynthesis of endogenous GSH via the activity of γ-glutamylcysteine synthase. The aim of this study is to investigate whether NAC supplementation can enhance the exercise training-induced improvements on physical fitness and metabolic health in adult men and women with overweight/obesity.

DETAILED DESCRIPTION:
Forty adults with overweight/obesity (both males and females, aged 35-45 years) who will meet the inclusion criteria will be randomly assigned to a Placebo (Pla, n=20, will be supplemented with 2 placebo pills daily over a 12-week period) or a NAC (NAC, n=20 will be supplemented with 2 pills x 600 mg N-acetylcysteine daily over a 12-week period) group. Both groups will participate in 3 multicomponent high-intensity interval training (m-HIIT) sessions per week over a 12-week period. At baseline, 6 weeks and 12 weeks participants will undergo assessment of their (i) anthropometrics (body weight, waist and hip circumferences) (ii) body composition (through total body DXA scan), (iii) fat liver content (via high-resolution ultrasound), (iv) cardiorespiratory fitness (determination of VO2max), (v) muscle strength (upper and lower body), (vi) habitual physical activity level (via accelerometry) and (vii) daily dietary intake (via dietary recalls). In addition, at the same time-points (Baseline, 6 weeks, 12 weeks), resting blood samples will be collected for the determination of (viii) blood redox status [reduced glutathione (GSH), oxidized glutathione (GSSH), GSH/GSSG, glutathione peroxidase (GPx), glutathione reductase (GR), superoxide dismutase (SOD) and catalase (CAT)], (ix) peripheral blood mononuclear cells antioxidant levels and markers of oxidative stress and inflammation (catalase, superoxide dismutase, glutathione peroxidase, glutathione reductase, malondialdehyde, TNF-α and Interleukin-6), (x) low-grade systemic inflammation [C-reactive protein (CRP) and Interleukin-6 (IL-6)], (xi) lipidemic profile (triglycerides, total cholesterol, HDL, LDL) and (xii) liver function (SGPT, SGOT, γ-GT, ALP, Fetuin-A), and (xiii) an oral glucose tolerance test (using 75g glucose loading) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-35 kg/m2
* Free of musculoskeletal injuries
* Free of chronic non-communicable diseases
* Do not receive any drug therapy
* Do not receive dietary supplements
* Normal menstrual cycle (for females)
* Non smokers

Exclusion Criteria:

* NAC intolerance
* Bleeding disorders
* Kidney disease
* Asthma
* Usage of blood thinners and/or angina medication

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight (kg) | At baseline, 6 weeks and 12 weeks
Change in waist circumference | At baseline, 6 weeks and 12 weeks
Change in hip circumference | At baseline, 6 weeks and 12 weeks
Change in fat mass (kg) | At baseline, 6 weeks and 12 weeks
  Fat mass will be assessed through dual energy X-ray absorptiometry (DXA)
Change in body fat percent (%) | At baseline, 6 weeks and 12 weeks
  Body fat percent will be assessed through dual energy X-ray absorptiometry (DXA)
Change in fat free mass (kg) | At baseline, 6 weeks and 12 weeks
  Fat free mass will be assessed through dual energy X-ray absorptiometry (DXA)
Change in lean body mass (kg) | At baseline, 6 weeks and 12 weeks
  Lean body mass will be assessed through dual energy X-ray absorptiometry (DXA)
Change in liver fat infiltration | At baseline and 12 weeks
  Liver fat infiltration will be assessed through ultrasound elastography
Change in cardiorespiratory fitness | At baseline, 6 weeks and 12 weeks
  Maximal oxygen consumption (VO2max) will be estimated during a single stage treadmill test (Ebbeling single stage test)
Change in lower body muscle strength | At baseline, 6 weeks and 12 weeks
  Maximal concentric peak torque will be assessed on an isokinetic dynamometer
Change in upper body muscle strength | At baseline, 6 weeks and 12 weeks
  Upper body muscle strength will be assessed through the abdominal strength test and the push-up test
Change in reduced glutathione (GSH) concentration | At baseline, 6 weeks and 12 weeks
  GSH concentration will be determined in blood erythrocytes and peripheral blood mononuclear cells
Change in oxidized glutathione (GSSG) concentration | At baseline, 6 weeks and 12 weeks
  GSSG concentration will be determined in blood erythrocytes and peripheral blood mononuclear cells
Change in glutathione peroxidase (GPx) activity | At baseline, 6 weeks and 12 weeks
  GPx activity will be determined in blood erythrocytes and peripheral blood mononuclear cells
Change in glutathione reductase (GR) activity | At baseline, 6 weeks and 12 weeks
  GR activity will be determined in blood erythrocytes and peripheral blood mononuclear cells
Change in catalase activity | At baseline, 6 weeks and 12 weeks
  Catalase activity will be determined in blood erythrocytes and peripheral blood mononuclear cells
Change in superoxide dismutase (SOD) activity | At baseline, 6 weeks and 12 weeks
  SOD activity will be determined in blood erythrocytes and peripheral blood mononuclear cells
Change in malondialdehyde concentration | At baseline, 6 weeks and 12 weeks
  Malondialdehyde concentration will be determined in peripheral blood mononuclear cells
Change in C-reactive protein (CRP) concentration | At baseline, 6 weeks and 12 weeks
Change in TNF-α concentration | At baseline, 6 weeks and 12 weeks
  TNF-α concentration will be determined in blood and peripheral blood mononuclear cells
Change in interleukin-6 (IL-6) concentration | At baseline, 6 weeks and 12 weeks
  IL-6 concentration will be determined in blood and peripheral blood mononuclear cells
Change in HDL cholesterol concentration | At baseline, 6 weeks and 12 weeks
  HDL cholesterol concentration will be determined in blood
Change in LDL cholesterol concentration | At baseline, 6 weeks and 12 weeks
  LDL cholesterol concentration will be determined in blood
Change in total cholesterol concentration | At baseline, 6 weeks and 12 weeks
  Total cholesterol concentration will be determined in blood
Change in triglycerides concentration | At baseline, 6 weeks and 12 weeks
  Triglycerides concentration will be determined in blood
Change in serum glutamic-oxaloacetic transaminase (SGOT/AST) concentration | At baseline, 6 weeks and 12 weeks
  SGOT concentration will be determined in blood
Alanine Aminotransferase (SGPT/ALT) concentration | At baseline, 6 weeks and 12 weeks
  SGPT concentration will be determined in blood
Change in Gamma-glutamyl transpeptidase (γ-GT) concentration | At baseline, 6 weeks and 12 weeks
  γ-GT concentration will be determined in blood
Change in fetuin-A concentration | At baseline, 6 weeks and 12 weeks
  Fetuin-A concentration will be determined in blood
Change in alkaline phosphatase (ALP) concentration | At baseline, 6 weeks and 12 weeks
  ALP concentration will be determined in blood
Change in glucose concentration | At baseline, 6 weeks and 12 weeks
  Glucose concentration will be determined in blood
Change in glycated hemoglobin (HbA1c) concentration | At baseline, 6 weeks and 12 weeks
  HbA1c concentration will be determined in blood
Change in insulin concentration | At baseline, 6 weeks and 12 weeks
  Insulin concentration will be determined in blood

SECONDARY OUTCOMES:
Change in dietary intake | At baseline, 6 weeks and 12 weeks
  Dietary intake will be monitored through diet recalls
Change in total number of steps | At baseline, 6 weeks and 12 weeks
  Total number of steps performed per day will be assessed by using accelerometers
Change in time spent in moderate-to-vigorous physical activity | At baseline, 6 weeks and 12 weeks
  The time spent in moderate-to-vigorous physical activity per day will be assessed by using accelerometers

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Rosvoglou, PhDc, Principal Investigator — University of Thessaly, Department of Physical Education and Sport Science; Dimitrios Draganidis, PhD, Study Director — University of Thessaly, Department of Physical Education and Sport Science
Locations (1):
- Department of Physical Education and Sport Science, University of Thessaly, Trikala, Karies, Greece